CLINICAL TRIAL: NCT04740918
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase III Study of the Efficacy and Safety of Trastuzumab Emtansine in Combination With Atezolizumab or Placebo in Patients With HER2-Positive and PD-L1-Positive Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Trastuzumab- (+/- Pertuzumab) and Taxane-Based Therapy (KATE3)
Brief Title: A Study of Trastuzumab Emtansine in Combination With Atezolizumab or Placebo as a Treatment for Participants With Human Epidermal Growth Factor 2 (HER2)-Positive and Programmed Death-ligand 1 (PD-L1)-Positive Locally Advanced (LABC) or Metastatic Breast Cancer (MBC)
Acronym: KATE3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to low enrollment, the Sponsor decided to prematurely terminate the study
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO42319; 2020-002818-41 (EudraCT Number)
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; atezolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Trastuzumab Emtansine and Placebo (Active Comparator): Placebo matched to atezolizumab followed by trastuzumab emtansine 3.6 milligrams per kilogram (mg/kg) intravenous (IV) infusion on Day 1 Cycle 1 and thereafter on Day 1 of each 21-day cycle until disease progression, unmanageable toxicity, or study termination by the sponsor.
  Interventions: Drug: Trastuzumab Emtansine; Other: Placebo
- Arm B: Trastuzumab Emtansine and Atezolizumab (Experimental): Atezolizumab 1200 mg IV infusion followed by trastuzumab emtansine 3.6 mg/kg IV infusion on Day 1 Cycle 1 and thereafter on Day 1 of each 21-day cycle until disease progression, unmanageable toxicity, or study termination by the Sponsor.
  Interventions: Drug: Trastuzumab Emtansine; Drug: Atezolizumab

INTERVENTIONS:
Drug: Trastuzumab Emtansine — Trastuzumab emtansine 3.6 mg/kg IV infusion
  Other Names: Kadcyla, T-DM1, RO5304020
Drug: Atezolizumab — Atezolizumab 1200 mg IV infusion
  Other Names: Tecentriq, RO5541267, MPDL3280A
  Arms: Arm B: Trastuzumab Emtansine and Atezolizumab
Other: Placebo — Placebo matched to atezolizumab
  Arms: Arm A: Trastuzumab Emtansine and Placebo

SUMMARY:
This study will evaluate the efficacy, safety and patient-reported outcomes of trastuzumab emtansine plus atezolizumab compared with trastuzumab emtansine plus placebo in participants with HER2-positive and PD-L1-positive LABC or MBC.Participants must have progressed either during or after prior trastuzumab- (+/- pertuzumab) and taxane-based therapy for LABC/MBC; or during (or within 6 months after completing) trastuzumab- (+/-pertuzumab) and taxane-based therapy in the neoadjuvant and/or adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* HER2+ and PD-L1+ locally advanced (LABC) or metastatic breast cancer (MBC)
* Progression must have occurred during most recent treatment for LABC/MBC or during, or within 6 months after completing, neoadjuvant and/or adjuvant therapy
* Prior treatment with trastuzumab (+/- pertuzumab) and taxane in the neoadjuvant and/or adjuvant, locally advanced, or metastatic setting
* No more than two prior lines of therapy in the metastatic setting
* Measurable disease per RESIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy >= 6 months
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Prior treatment with trastuzumab emtansine in metastatic setting
* History of exposure to cumulative doses of anthracyclines
* Symptomatic or actively progressing central nervous system (CNS) metastases; asymptomatic CNS lesions ≤ 2cm without clinical requirement for local intervention or asymptomatic patients with treated CNS lesions are eligible
* Current Grade >= 3 peripheral neuropathy
* Cardiopulmonary dysfunction
* History of malignancy within 5 years prior to initiation of study treatment, with the exception of the cancer under investigation and malignancies with a negligible risk of metastasis or death
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* Active hepatitis B, hepatitis C and/or tuberculosis
* Prior allogeneic stem cell or solid organ transplantation
* Receipt of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, during treatment, or within 5 months following the last dose of study treatment
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- Emad Ibrahim, Md, Inc, Redlands, California, United States
- Peter MacCallum Cancer Center, Melbourne, Victoria, Australia
- Brazil (5):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo, São Paulo
- Canada (2):
  - Royal Victoria Hospital, Barrie, Ontario
  - Centre Hospitalier de l?Université de Montréal (CHUM), Montreal, Quebec
- China (10):
  - Peking University People's Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- Colombia (2):
  - Clinica Vida, Medellín
  - Oncomedica S.A., Montería
- Croatia (2):
  - Clinical Hospital Center Sestre Milosrdnice, Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Institut Curie - Hopital Rene Huguenin, Saint-Cloud, France
- Italy (3):
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino, Campania
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE, Napoli, Campania
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna, Emilia-Romagna
- Oslo Universitetssykehus HF, Oslo, Norway
- Philippines (3):
  - Cebu Doctors' University Hospital, Cebu City
  - St. Luke's Medical Center, Quezon City
  - Cardinal Santos Medical Center, San Juan City
- Poland (2):
  - Opolskie Centrum Onkologii, Opole
  - Centrum Onkologii ? Instytut im. Marii Sk?odowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- Portugal (2):
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
  - IPO do Porto, Porto
- SBIH Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa, Bashkortostan Republic, Russia
- Seoul National University Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario La Paz, Madrid
- Turkey (Türkiye) (7):
  - Adana Baskent University Medical Faculty, Adana
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi, Adapazari/Sakarya
  - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul
  - Acibadem University School of Medicine Altunizade Hospital Oncology Service, Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Kayseri Acibadem Hospital, Kayseri
  - Hacettepe Uni Medical Faculty Hospital, Sihhiye/Ankara
- United Kingdom (3):
  - UCL Hospital NHS Trust, London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Nottingham University Hospitals City Campus, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 96 participants with human epidermal growth factor receptor 2 (HER2)-positive and programmed death-ligand 1 (PD-L1)-positive locally advanced (LABC) or metastatic breast cancer (MBC) took part in the study across 52 investigative sites in 19 countries from 07 June 2021 to 19 June 2024.
Pre-assignment Details: Participants were randomized in 1:1 ratio to receive trastuzumab emtansine + placebo or trastuzumab emtansine + atezolizumab.
Groups:
- Trastuzumab Emtansine 3.6 mg + Placebo: Participants received trastuzumab emtansine, 3.6 milligrams (mg), every 3 weeks (Q3W) as an intravenous (IV) infusion in combination with atezolizumab matching placebo, Q3W as an IV infusion on Day 1 of each 21-day cycle until radiographic disease progression, intolerable toxicity, withdrawal of consent, death or study termination by the sponsor.
- Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg: Participants received trastuzumab emtansine, 3.6 mg, Q3W as an IV infusion in combination with atezolizumab, 1200 mg, Q3W as an IV infusion on Day 1 of each 21-day cycle until radiographic disease progression, intolerable toxicity, withdrawal of consent, death or study termination by the sponsor.
Period: Overall Study
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Started | 50 | 46
Safety Population (Safety evaluable population included all participants who received at least one full or partial dose of study drug. 1 participant randomized to Trastuzumab Emtansine + Placebo moved to Trastuzumab Emtansine + Atezolizumab 1200 mg. Hence, has been represented in the later arm for safety analysis.) | 49 | 47
ITT With Brain Metastases (ITT with brain metastasis population included all participants in ITT with brain metastasis at randomization.) | 5 | 4
ITT With CNS Metastases (ITT with CNS metastasis population included all participants in ITT with CNS metastasis at randomization.) | 7 | 4
ITT Without CNS Metastases (ITT without CNS metastases population included all participants in the ITT without CNS metastasis at baseline.) | 43 | 42
ITT With Measurable Disease (ITT with measurable disease population included all participants in the ITT without CNS metastasis at baseline.) | 49 | 45
Completed | 0 | 0
Not Completed | 50 | 46
Not completed — Study Terminated by Sponsor | 41 | 32
Not completed — Death | 3 | 6
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Progressive disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all participants who were randomized in the study, whether or not they received any study medication.
Groups:
- Trastuzumab Emtansine 3.6 mg + Placebo: Participants received trastuzumab emtansine, 3.6 mg, Q3W as an IV infusion in combination with atezolizumab matching placebo, Q3W as an IV infusion on Day 1 of each 21-day cycle until radiographic disease progression, intolerable toxicity, withdrawal of consent, death or study termination by the sponsor.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.7) | 50.9 (10.0) | 52.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 46 | 96
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 42 | 39 | 81
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 17 | 21 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 29 | 23 | 52
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS was defined as the time from randomization to the first occurrence of documented disease progression (PD), as determined by the investigator according to RECIST v1.1 or death from any cause whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). Median PFS was calculated using the Kaplan-Meier (KM) methodology. Data for participants without PD or death from any cause as of the data cut-off date were censored at the time of the last tumor assessment.
Time Frame: Up to 28 months
Population: ITT population included all participants who were randomized in the study, whether they received any study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 50 | 46
months | 7.52 [6.18 to 10.94] | 8.61 [5.72 to 16.92]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — Cox proportional hazards model, stratified by local hormonal status (estrogen receptors (ER) and/or progesterone receptor (PgR) positive vs. ER and PgR negative/unknown) and Disease status (visceral metastasis without brain metastasis vs. non-visceral metastasis only without brain metastasis [including locally advanced disease] vs. Brain metastasis) were used to estimate the Hazard Ratio (HR); p = 0.2876, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.44 to 1.28]

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study treatment to the time of death from any cause. Participants who are alive as of the data cut-off date of the analysis were censored at the last known date they were alive. Participants with no post-baseline information were censored at the date of randomization plus 1 day. Median OS was calculated using the KM methodology.
Time Frame: Up to 28 months
Population: ITT population included all participants who were randomized in the study, whether they received any study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 50 | 46
months | NA [NA to NA] — The median and 95% confidence interval (CI) was not estimable due to insufficient number of events. | NA [21.29 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — Cox proportional hazards model, stratified by local hormonal status (ER and/or PgR positive vs. ER and PgR negative/unknown) and Disease status (visceral metastasis without brain metastasis vs. non-visceral metastasis only without brain metastasis [including locally advanced disease] vs. Brain metastasis) were used to estimate the HR; p = 0.5151, Log Rank; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [0.39 to 6.43]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with complete response (CR) or partial response (PR) on two consecutive assessments, at least 28 days apart, as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. Only participants with measurable disease at baseline were analyzed for this outcome measure. Participants without a post-baseline tumor assessment were considered non-responders. An estimate of the ORR and its 95% CI (Wilson score confidence interval) were calculated for each treatment arm.
Time Frame: Up to 28 months
Population: Subset ITT with measurable disease included all participants in the ITT with a measurable disease at baseline. ITT population included all participants who were randomized to the study, whether or not they received any study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 49 | 45
percentage of participants | 49 [34.64 to 63.48] | 53.3 [38.04 to 68.07]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — A Cochran-Mantel-Haenszel chi-square test, stratified by local hormonal status (ER and/or PgR positive vs. ER and PgR negative/unknown) and Disease status (visceral metastasis without brain metastasis vs. non-visceral metastasis only without brain metastasis [including locally advanced disease] vs. Brain metastasis), was used to test for difference in response rates; p = 0.7240, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.50 to 2.70]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was calculated for participants who had a best OR of CR/PR. DOR was defined as time from first occurrence of a documented OR until the time of documented PD or death from any cause, whichever occurs first as determined by investigator assessment using RECIST v1.1. CR=the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR=at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD=at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Median DOR was calculated using the KM methodology.
Time Frame: Up to 28 months
Population: Subset ITT with measurable disease included all participants in the ITT with a measurable disease at baseline. ITT population included all participants who were randomized to the study, whether or not they received any study medication. Overall number analyzed is the number of participants with OR, i.e, responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 24 | 24
months | 8.21 [5.72 to NA] — The upper limit of 95%CI was not estimable due to insufficient number of events. | 15.57 [7.06 to NA] — The upper limit of 95%CI was not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3531, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.26 to 1.61]

5. Secondary Outcome: PFS in Participants With Baseline Brain Metastases as Determined by Investigator Assessment Using RECIST v1.1
Description: PFS was defined as the time from randomization to the first occurrence of documented PD, as determined by the investigator according to RECIST v1.1 or death from any cause whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Median PFS was calculated using the KM methodology.
Time Frame: Up to 28 months
Population: ITT with brain metastasis population included all participants in ITT with brain metastasis at randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 5 | 4
months | 7.69 [4.14 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | 4.78 [1.31 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7175, Log Rank; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.27 to 6.81]

6. Secondary Outcome: OS in Participants With Baseline Brain Metastases
Description: OS is defined as the time from the first dose of study treatment to the time of death from any cause. Median OS was calculated using the KM methodology.
Time Frame: Up to 28 months
Population: ITT with brain metastasis population included all participants in ITT with brain metastasis at randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 5 | 4
months | NA [NA to NA] — The median and 95%CI was not estimable due to insufficient number of events. | NA [9.53 to NA] — The median and upper limit of 95%CI was not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3173, Log Rank

7. Secondary Outcome: Central Nervous System (CNS) PFS as Determined by Investigator Using RECIST v1.1 in Participants With Baseline CNS Metastases
Description: CNS PFS was defined as the time from randomization to the first occurrence of documented CNS PD, or first occurrence of symptomatic CNS disease as determined by the investigator according to RECIST v1.1 or death from any cause whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Median PFS was calculated using the KM methodology. Participants who experienced non-CNS PD at the time of analysis were censored at the date of this progression. Participants who experienced no PD and were alive at the time of analysis were censored at date of their last post-baseline tumor assessment or, if they had no post-baseline tumor assessment, on the date of randomization + 1 day.
Time Frame: Up to 28 months
Population: ITT with CNS metastasis population included all participants in ITT with CNS metastasis at randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 7 | 4
months | 10.41 [4.11 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | 9.53 [1.31 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.8658, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.16 to 8.60]

8. Secondary Outcome: CNS PFS as Determined by Investigator Using RECIST v1.1 in Participants Without Baseline CNS Metastases
Description: as for outcome 7
Time Frame: Up to 28 months
Population: ITT without CNS metastases at baseline population included all participants in the ITT without CNS metastasis at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 43 | 42
months | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of events. | NA [21.29 to NA] — The median and upper limit of 95% CI were not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine 3.6 mg + Placebo vs Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.8407, Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.27 to 4.99]

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: Up to 28 months
Population: Safety evaluable population included all participants who received at least one full or partial dose of study drug. One participant randomized to Trastuzumab Emtansine + Placebo moved to Trastuzumab Emtansine + Atezolizumab 1200 mg. Hence, has been represented in the later arm for safety analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 49 | 47
percentage of participants | 93.9 | 97.9

10. Other Pre Specified Outcome: PFS as Determined by a Blinded Independent Central Review (BICR) Committee Using RECIST v1.1
Description: PFS was defined as the time from randomization to the first occurrence of documented PD, as determined by the BICR committee according to RECIST v1.1 or death from any cause whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 28 months
Population: As prespecified in the latest protocol, following sponsor's decision to prematurely terminate the study, analysis of PFS as determined by a BICR committee was not conducted.
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Mean Absolute Scores in Physical Function (PF), Role Function (RF) and Global Health Status (GHS/QoL) Scores Measured Using European Organization for Research and Treatment of Cancer (EORTC QLQ-C30)
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The PF scale has 5 questions about participant's PF and daily activities (strenuous activities, long walks, short walks, bed/chair rest & needing help with eating, dressing, washing themselves, or using the toilet). The RF scale has 2 questions about work/daily activities and hobbies/leisurely activities. The PF and RF are scored on a 4-point scale (1=Not at All to 4=Very Much). The GHS/QoL are scored on a 7-point scale (1=Very Poor to 7=Excellent). The obtained scores are linearly transformed to a score range of 0-100, where higher scores indicate a higher response level and better QoL, functioning/support.
Time Frame: Up to 28 months
Population: As prespecified in the latest protocol, following sponsor's decision to prematurely terminate the study, the analysis for EORTC QLQ-C30 was not conducted.
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Change From-Baseline in PF, RF and GHS/QoL Scores Measured Using EORTC QLQ-C30
Description: as for outcome 11
Time Frame: Up to 28 months
Population: as for outcome 11
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Percentage of Participants With Clinically Meaningful Deterioration in PF, RF and GHS/QoL Measured Using EORTC QLQ-C30
Description: as for outcome 11
Time Frame: Up to 28 months
Population: as for outcome 11
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Maximum Serum Concentration (Cmax) of Trastuzumab Emtansine
Description: As prespecified in the latest protocol, following sponsor's decision to prematurely terminate the study, PK objectives and outcome measures were no longer applicable. Hence sample collection was stopped, and this outcome measure was not assessed or analyzed.
Time Frame: Up to 28 months
Population: As prespecified in the latest protocol, following sponsor's decision to prematurely terminate the study, PK objectives and outcome measures were no longer applicable. Hence sample collection was stopped, and this outcome measure was not assessed or analyzed.
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Cmax of Atezolizumab
Description: as for outcome 14
Time Frame: Up to 28 months
Population: as for outcome 14
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Trastuzumab Emtansine
Description: As prespecified in the latest protocol, following sponsor's decision to prematurely terminate the study, immunogenicity objectives and outcome measures were no longer applicable.
Time Frame: Up to 28 months
Population: As prespecified in the latest protocol, following sponsor's decision to prematurely terminate the study, immunogenicity objectives and outcome measures were no longer applicable.
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Percentage of Participants With ADAs to Atezolizumab
Description: as for outcome 16
Time Frame: Up to 28 months
Population: as for outcome 16
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 months
Description: Safety evaluable population included all participants who received at least one full or partial dose of study drug. One participant randomized to Trastuzumab Emtansine + Placebo moved to Trastuzumab Emtansine + Atezolizumab 1200 mg. Hence, has been represented in the later arm for safety analysis.
Arm/Group | Trastuzumab Emtansine 3.6 mg + Placebo | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg
All-Cause Mortality (participants affected / at risk) | 3/49 | 6/47
Serious Adverse Events (participants affected / at risk) | 9/49 | 14/47
Other Adverse Events (participants affected / at risk) | 46/49 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine 3.6 mg + Placebo (N=49) | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg (N=47)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine 3.6 mg + Placebo (N=49) | Trastuzumab Emtansine 3.6 mg + Atezolizumab 1200 mg (N=47)
Anaemia (Blood and lymphatic system disorders) | 10 (19) | 20 (36)
Leukopenia (Blood and lymphatic system disorders) | 3 (6) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (8) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (21) | 12 (20)
Hypothyroidism (Endocrine disorders) | 2 (2) | 7 (9)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (4)
Constipation (Gastrointestinal disorders) | 4 (6) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (15)
Nausea (Gastrointestinal disorders) | 12 (18) | 16 (30)
Vomiting (Gastrointestinal disorders) | 9 (16) | 8 (17)
Asthenia (General disorders) | 4 (7) | 7 (9)
Fatigue (General disorders) | 11 (15) | 11 (16)
Influenza like illness (General disorders) | 3 (4) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 3 (4) | 11 (16)
COVID-19 (Infections and infestations) | 4 (4) | 4 (5)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (6) | 3 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Alanine aminotransferase increased (Investigations) | 15 (25) | 23 (52)
Amylase increased (Investigations) | 0 (0) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 23 (33) | 26 (52)
Blood alkaline phosphatase increased (Investigations) | 4 (9) | 11 (19)
Blood bilirubin increased (Investigations) | 2 (5) | 7 (23)
Blood cholesterol increased (Investigations) | 1 (1) | 3 (5)
Blood lactate dehydrogenase increased (Investigations) | 8 (14) | 11 (19)
Gamma-glutamyltransferase increased (Investigations) | 6 (8) | 11 (15)
Lipase increased (Investigations) | 0 (0) | 6 (8)
Lymphocyte count decreased (Investigations) | 2 (2) | 5 (16)
Neutrophil count decreased (Investigations) | 2 (2) | 10 (28)
Platelet count decreased (Investigations) | 11 (21) | 18 (40)
Weight decreased (Investigations) | 3 (3) | 5 (6)
White blood cell count decreased (Investigations) | 2 (3) | 7 (32)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 14 (40)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 6 (15)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 3 (5) | 2 (2)
Headache (Nervous system disorders) | 8 (17) | 9 (12)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 6 (6)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (6) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
The Sponsor decided to prematurely terminate the study due to a lower-than-expected enrollment rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT04740918/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT04740918/SAP_001.pdf